CLINICAL TRIAL: NCT02735837
Title: The Effect of Non-Surgical Periodontal Therapy With Adjunctive Topical Doxycycline Gel on HbA1c in Patients With Type 2 Diabetes Mellitus (DM):A Randomized, Clinical Trial
Brief Title: The Effect of Topical Doxycycline Gel on HbA1c in Patients With Type 2 Diabetes Mellitus(DM) ®
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Amirhossein Farahmand (Other)
Responsible Party: Sponsor-Investigator, Amirhossein Farahmand, The effect of non-surgical periodontal therapy with adjunctive topical doxycycline gel on HbA1c in patients with type 2 diabetes mellitus (DM)., Islamic Azad University, Sanandaj
Organization: Islamic Azad University, Sanandaj (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 560
Record Dates: First submitted 2016-03-30; First posted 2016-04-13 (Estimated); Last update posted 2019-07-05 (Actual); Status verified 2019-07

CONDITIONS: Diabetes Mellitus With Periodontal Disease
MeSH Terms: interventions — Doxycycline; Gels

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- doxycycline gel (Active Comparator): Doxycycline 3% topical gel was put into the periodontal pocket using an insulin syringe
  Interventions: Drug: Doxycycline Group
- placebo gel (Placebo Comparator): placebo topical gel was put into the periodontal pocket using an insulin syringe
  Interventions: Drug: placebo topical gel

INTERVENTIONS:
Drug: Doxycycline Group — Doxycycline 3% topical gel was put into the periodontal pocket using an insulin syringe
  Other Names: Doxycycline 3% topical gel; Group A
  Arms: doxycycline gel
Drug: placebo topical gel — placebo topical gel was put into the periodontal pocket using an insulin syringe
  Other Names: Group B
  Arms: placebo gel

SUMMARY:
Aim:

The purpose of this study is to investigate the effect of nonsurgical periodontal therapy plus subgingivally doxycycline gel 3% on glycemic control in type 2 diabetes mellitus (type 2 DM) patients who have periodontitis.

Materials and methods:

A total of 24 type 2 DM patients with periodontitis will be selected for the study, and randomly divided into two equal groups,who are at least 35 years of age and 16 teeth and type II diabetes are (at least the last 3 months of diagnosis of diabetes and its FBS More than 110 have), and also with periodontal disease are chronic moderate (at least in three areas Attachment level to a depth of 3-4 mm maxillary or mandibular been confirmed by clinical examination and radiographic signs are being); Takes place. The initial HbA1c Patients should be between 7-9 percent over the past three months has changed his medication also found the necessary explanations on how to do that consent, Plaque index (PI) by Loe & Silness, bleeding on probing (BOP) based on Carter and Barnes (if any bleeding number 1 and its absence is 0), probing depth (PD) and clinical attachment levels (CAL) were recorded. "Group 1": (12 patients) was treated with oral hygiene instruction, scaling and root planing, and doxycycline gel for 15 days; and "Group 2": (12 patients) has the same treatment but with placebo gel, After 12 weeks their periodontal condition and Fasting blood sugar (FBS), glycated hemoglobin (HbA1c) level, will be reevaluated.

DETAILED DESCRIPTION:
Doxycycline downregulates the activity of matrix metalloproteinases (MMPs), key destructive enzymes in periodontal disease

ELIGIBILITY:
Inclusion Criteria:

* Patients with diabetes mellitus type II (at least 3 months before diagnosis, and A fasting blood sugar level of more than 125 mg/dl) and has periodontal disease is a chronic moderate (has a clinical attachment level of 3-4 mm) peritonitis
* Minimum of 16 natural teeth, and no periodontal treatment in the prior 6 months, - Had a glycated α hemoglobin (HbA1c) value between 7- 9 percent at screening
* Had reported no changes in diabetes medications within the last 3 months were in the care of a physician for their diabetes.

Exclusion Criteria:

* Pregnancy or lactation
* History of allergy to drugs used in the study
* Smoking
* Diabetes-related emergency within 30 days ago
* Use of nonsteroidal anti-inflammatory drugs
* Or taking low dose daily aspirin (75-325 mg)\
* Use of immunosuppressive medications; antibiotic use
* Dialysis
* Risk of bleeding complications
* The type of disease periodontal (Aggressive)
* A history of periodontal treatment in the previous 6 months
* Orthodontic treatment
* Using the removal prostheses
* Extensive dental caries
* Dental abscesses or infections.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2015-01; Primary Completion 2016-03 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Periodontal pocket | 15 days
  Periodontal probe

SECONDARY OUTCOMES:
glycated hemoglobin (HbA1c) | 3 months
  Blood test

IPD SHARING:
Plan to Share IPD: Yes